CLINICAL TRIAL: NCT00839280
Title: Evaluation of the Moisturizing Effect of Bepanthen Burn Relief Foam Spray New Formula Versus Bepanthen Burn Relief Foam Spray (Current Formula). Equivalence Trial. Intra-individual Design.
Brief Title: Moisturizing Effect of Two Dexpanthenol Formulations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12040
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Skin Abnormalities
Keywords: Dry skin; Dexpanthenol; Moisturizing effect
MeSH Terms: conditions — Skin Abnormalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Dexpanthenol foam spray, new formulation
- Arm 2 (Active Comparator)
  Interventions: Drug: Dexpanthenol foam spray, old formulation

INTERVENTIONS:
Drug: Dexpanthenol foam spray, new formulation — 2 applications of 2 micro liter/square centimeter on a 4X4 cm area corresponding to 32 micro liter
  Arms: Arm 1
Drug: Dexpanthenol foam spray, old formulation — 2 applications of 2 micro liter/square centimeter on a 4X4 cm area corresponding to 32 micro liter
  Arms: Arm 2

SUMMARY:
The study focuses to prove the equivalent moisturizing effect of two different Dexpanthenol formulations

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Phototype: I to IV according to Fitzpatrick scale
* Subjects with dry skin on their forearms

Exclusion Criteria:

* Pregnant or nursing women
* Subjects registered as being in exclusion period in the French Health Minister file of subjects
* Subjects with hypersensitivity to one of the test products

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2007-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) of the cutaneous hydration rate measured with corneometer between T0 and T5h | 0 min, 15 min, 30 min, 1h, 2h, 3h, 5h

SECONDARY OUTCOMES:
Cutaneous hydration rate | 15 min, 30 min, 1h, 2h, 3h, 5h
Incidence of Adverse Events | FPFV - LPLV

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Villeurbanne, France